CLINICAL TRIAL: NCT01306240
Title: Surfactant Treatment Compared to Nasal Continuous Positive Airway Pressure for the Management of Respiratory Distress Syndrome in the Newborn Between 35 and 41 Weeks of Gestation
Brief Title: Surfactant Versus Nasal Continuous Positive Airway Pressure (nCPAP) for Respiratory Distress Syndrome in the Newborn ≥ 35 Weeks of Gestation
Acronym: ASPEN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruiting problems
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHRCIR09-DR-TOURNEUX
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Infant newborn; Infant preterm; Acute respiratory distress syndrome; surfactant; Hyaline Membrane disease; Newborn acute respiratory distress syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome; Hyaline Membrane Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early strategy (Experimental): Intratracheal poractant alpha (Curosurf®) after tracheal intubation
  Interventions: Procedure: Surfactant instillation
- Delayed strategy (Active Comparator): Nasal Continous Positive Airways Pressure. Intratracheal poractant alpha as a rescue treatment if FiO2 > 60%
  Interventions: Procedure: nCPAP

INTERVENTIONS:
Procedure: Surfactant instillation — Intra-tracheal poractant alpha instillation after tracheal intubation
  Arms: Early strategy
Procedure: nCPAP — Nasal Continous Positive Airways Pressure (nCPAP). Positive End Expiratory Pressure (PEEP) is set between 4 to 6 cm H2O. FiO2 is adjusted for a target post-ductus arteriosus SpO2 between 92% and 96%.
  Arms: Delayed strategy

SUMMARY:
Term and near term newborns can present acute respiratory distress syndrome (RDS). Surfactant treatment has been shown effective in reducing mechanical ventilation and oxygen treatment durations in the preterm newborn. Whether surfactant treatment is beneficial for term and near term newborns is unknown. The purpose of this study is to compare surfactant treatment vs. nasal continuous positive airways pressure in the newborn between 35 and 41 weeks of gestation with RDS within the first 24 hours of life. The study's primary endpoint is "survival with no oxygen treatment at 72 hours of life". The secondary endpoints are: death, surfactant treatment, pneumothorax, secondary infections, pulmonary hypertension, inhaled nitric oxide treatment, fluid loading treatment, vasopressive amines treatment, mechanical ventilation duration, nCPAP treatment duration, Oxygen treatment duration, Oxygen treatment at 28 days of life, hospitalization duration and treatment strategy cost.

DETAILED DESCRIPTION:
Newborn between 35 and 41 weeks of gestation with RDS within the first 24 hours of life, treated with nCPAP and a FiO2 ≥ 30% are eligible. Randomisation is stratified by centre and 2 age groups (35-36 weeks of gestation and 37-41 weeks ogf gestation). One arm will receive surfactant treatment after tracheal intubation. The second arm will continue nCPAP. A rescue treatment is used in the second arm if FiO2 > 60%. In each arm the newborn is weaned from mechanical ventilation and oxygen treatment as soon as possible. The primary outcome of the study is the success of the procedure defined as "survival without any oxygen treatment" at 72 hours of life.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 35 and 41 weeks of gestation
* < 24 hours of life
* Nasal Continuous Positive Airways Pressure (nCPAP) for more than 1 hour
* FiO2 ≥ 30% with nCPAP and a target post-ductus arteriosus SpO2 >92%
* Written consent of the parents

Exclusion Criteria:

* FiO2 > 60% with nCPAP, ou FiO2 > 40% for 3 consecutives hours whatever the respiratory support
* Life threatening congenital pathology
* Congenital cardiopathy (except patent ductus arteriosus)
* Shock defined as systemic hypotension (mean blood pressure <10th percentile of the normal range for birth weight and postnatal age) with at least 3 of the following criteria for decrease perfusion: 1) tachycardia (heart rate > 160 beats/min); 2) abnormal peripheral pulses; 3) modified extremities coloration; 4) prolonged capillary refill time > 3 seconds; 5) urine output < 1 ml/kg/h
* Blood gas pH < 7.19 and / or PCO2 > 65 mmHg
* Apgar score ≤ 3 at 5 minutes of life

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Succes of the procedure | 72 hours of life
  survival without any oxygen treatment

SECONDARY OUTCOMES:
Morbidity associated to the management of a newborn with RDS in a neonatal intensive care unit | Every 8 hours of life between birth and 72 hours of life. Then every day until neonatal intensive care unit discharge.
  * Death
  * Surfactant treatment,
  * Pneumothorax,
  * Secondary infections,
  * Pulmonary hypertension,
  * Inhaled nitric oxide treatment,
  * Fluid loading treatment,
  * Vasopressive amines treatment,
  * Mechanical ventilation duration,
  * nCPAP treatment duration,
  * Oxygen treatment duration,
  * Oxygen treatment at 28 days of life
  * Hospitalization duration
  * Treatment strategy cost

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens University Hospital, Amiens, Picardie, France